CLINICAL TRIAL: NCT05164341
Title: A 12-Month Randomized, Multicenter, Double-Blind, Placebo-Controlled Phase 3 Study to Evaluate the Safety and Efficacy of Daily Subcutaneous Metreleptin Treatment in Subjects With Partial Lipodystrophy
Brief Title: Study to Evaluate the Safety and Efficacy of Daily Subcutaneous Metreleptin Treatment in Subjects With PL
Acronym: METRE-PL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amryt Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APG-20
Record Dates: First submitted 2021-11-11; First posted 2021-12-20 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Partial Lipodystrophy
Keywords: metreleptin
MeSH Terms: conditions — Lipodystrophy, Partial, Acquired | interventions — metreleptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- metreleptin (Active Comparator): Metreleptin [Recombinant-methionyl human Leptin; r-metHuLeptin] for daily injection is a sterile, white, solid lyophilised cake
  Interventions: Drug: metreleptin
- placebo (Placebo Comparator): Placebo for daily injection is a sterile, white, solid lyophilised cake
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: metreleptin — Metreleptin is a recombinant human leptin analog that is indicated as an adjunct to diet as replacement therapy to treat the complications of leptin deficiency
  Arms: metreleptin
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
This is a Phase III, double-blind, placebo-controlled, safety and efficacy study of daily SC metreleptin in subjects with Partial Lipodystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Familial Partial Lipodystrophy (FPLD)
* Subjects with poor metabolic control defined as:

HbA1c ≥7% (at Visit 1 and Visit 3) and/or Fasting TGs ≥500 mg/dL (5.65 mmol/L, at Visit 1 and Visit 3)

* Patients should be receiving optimized stable therapy

Exclusion Criteria:

* Previous treatment with metreleptin
* Leptin levels >20.0 ng/mL
* Acquired or radiation induced partial lipodystrophy (APL)

Other protocol defined inclusion/exclusion criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to month 6 in HbA1c in subjects with partial lipodystrophy (PL) | 6 months
  To evaluate the efficacy (HbAa1c) of daily SC metreleptin treatment
Percent change from Baseline to month 6 in fasting TGs in subjects with partial lipodystrophy (PL) | 6 months
  To evaluate the efficacy (TGs) of daily SC metreleptin treatment

SECONDARY OUTCOMES:
Safety analysis of AEs, AESIs, SAEs by treatment arm | 12 months
  To evaluate the safety of daily SC metreleptin treatment in subjects with PL
Change from baseline to months 9 and 12 in HbA1c in subjects with partial lipodystrophy (PL) | 12 months
  To assess the effect of metreleptin on HbA1c
Percent change from baseline to months 9 and 12 in fasting TGs in subjects with partial lipodystrophy (PL) | 12 months
  To assess the effect of metreleptin on TGs
Change from Baseline to each assessment time point in quality of life (QoL) in all subjects | 12 months
  To assess the effect of metreleptin on quality of life (QoL) in all subjects

CONTACTS AND LOCATIONS:
Locations (31):
- United States (13):
  - University of Alabama, Birmingham, Alabama
  - UC Davis, Sacramento, California
  - Flourish Boca Raton, Boca Raton, Florida
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - Amryt Research Site, Endocrinology Research Associates Inc, Columbus, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- UZ Leuven, Leuven, Belgium
- Brazil (4):
  - Universitário Walter Cantídio, Fortaleza
  - Insight Centro de Pesquisas, Porto Alegre
  - Hospital das Clinicas FMRP-USP, Ribeirão Preto
  - Instituto Estadual de Diabetes e Endocrinologia (IEDE-RJ), Rio de Janeiro
- Canada (6):
  - Nova Scotia Health, Halifax, Nova Scotia
  - Care Access Clinic, Sydney, Nova Scotia
  - Hamilton General Hospital- McMaster University, Hamilton, Ontario
  - London Health Science Centre, London, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Faculty of Medicine, Universite Laval, Québec, Quebec
- Universidad Catolica, Santiago, Chile
- Hadassah University Hospital - Ein Kerem, Jerusalem, Israel
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Radboud University Medical Centre Interne Geneeskund, Nijmegen
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Katowice
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
- University Clinical Hospital of Santiago de Compostela/Hospital Universitario, Santiago de Compostela, Spain